CLINICAL TRIAL: NCT03059927
Title: The Effect of Three Prosthesis Designs on Implant Stability and Survival, Knee Function, and Clinical Course in Knee Arthroplasty: a Randomized Trial
Brief Title: The Effect of Three Prosthesis Designs in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lovisenberg Diakonale Hospital (Other)
Collaborators: Haugesund Rheumatism Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LovisenbergOrto
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-02

CONDITIONS: Gonarthrosis; Primary; Degenerative Joint Disease of Knee
Keywords: Cruciate retaining; Anterior stabilized; Posterior stabilized; Posterior cruciate ligament; Degenerative knee joint disease; Knee injury and Osteoarthritis Outcome Score; Kinematic radiostereometry
MeSH Terms: conditions — Osteoarthritis, Knee; Knee Injuries | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Knee arthroplasty, Cruciate retaining (Active Comparator): Total knee replacement with preserved posterior cruciate ligament and a cruciate retaining insert.
  Interventions: Procedure: Knee arthroplasty, Cruciate retaining
- Knee arthroplasty, Anterior stabilized (Active Comparator): Total knee replacement with sacrificed posterior cruciate ligament and an anterior stabilized insert.
  Interventions: Procedure: Knee arthroplasty, Anterior stabilized
- Knee arthroplasty, Posterior stabilized (Active Comparator): Total knee replacement with sacrificed posterior cruciate ligament and a posterior stabilized design.
  Interventions: Procedure: Knee arthroplasty, Posterior stabilized

INTERVENTIONS:
Procedure: Knee arthroplasty, Cruciate retaining — Legion total knee arthroplasty implant component, Smith & Nephew, Cruciate Retaining design
  Arms: Knee arthroplasty, Cruciate retaining
Procedure: Knee arthroplasty, Anterior stabilized — Legion total knee arthroplasty implant component, Smith & Nephew, Anterior Stabilized design
  Arms: Knee arthroplasty, Anterior stabilized
Procedure: Knee arthroplasty, Posterior stabilized — Legion total knee arthroplasty implant component, Smith & Nephew, Posterior Stabilized design
  Arms: Knee arthroplasty, Posterior stabilized

SUMMARY:
The purpose of this study is to compare three prosthesis designs to compare three prosthesis designs for total knee arthroplasty and determine the best option for patients in need of a knee replacement.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is a cost beneficial surgery shown to improve pain, function and quality of life in patients with osteoarthritis. In 2015, 6093 patients received primary TKA in Norway. Despite the procedure´s general success, 20% of patients report persistent postoperative pain and/or dissatisfaction with the surgical outcome. Efforts to further improve the procedure have raised considerable debate regarding the role and management of the posterior cruciate ligament (PCL). Prostheses for TKA have evolved into designs that either preserve or sacrifice the PCL. In patients with a functional PCL, the decision of which design is selected depends largely on the favor and training of the surgeon. To further improve TKA patient outcomes, a better understanding of the role of these differing PCL treatments is needed. Thus, the aim of this study is to determine whether patients' perceived outcome, implant stability and clinical outcome differ between 3 TKA implant designs (2 PCL-sacrificing and 1 PCL-retaining). We will conduct a 3-arm randomized controlled prospective trial with 5-year follow-up. This study will have impact on clinical practice by addressing the lack of evidence supporting use of these different types of implants.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis
* Non-fixed or fixed varus or valgus deformity less than 15º measured on preoperative standing hip-knee-ankle (HKA) radiographs
* Intact PCL (assessed preoperatively and verified during surgery)
* Age 45 - 75 years (only patients 45 - 70 years will be included in the kinematic RSA)
* Body mass index ≤ 35 kg/m2
* ASA (American Society of Anaesthesiologists) score I or II
* Only patients with KOOS scores above 80 on the Symptoms, ADL (Activities of Daily Living) and Pain subscales will be included in the kinematic analysis

Exclusion Criteria:

* Prior ACL (anterior cruciate ligament) surgery
* Impaired collateral ligaments
* Secondary osteoarthritis of the knee
* Previous osteotomy
* Rheumatic disease
* Flexion less than 90 degrees
* Flexion contracture over 10 degrees
* Peripheral neuropathy
* Malignancy
* Patients who do not speak Norwegian

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee injury and osteoarthritis outcome score (KOOS) | Pre-operative, 1, 2 and 5 years
  KOOS is a knee-specific questionnaire developed to evaluate short- and long-term symptoms and functioning in subjects with knee injury and osteoarthritis. KOOS is validated for use in total knee arthroplasty and has been shown to be a valid, reliable and responsive measure. KOOS is a patient-administered questionnaire.

SECONDARY OUTCOMES:
Oxford knee score (OKS) | Pre-operative, 1, 2 and 5 years
  OKS is a brief patient-completed questionnaire for patients undergoing total knee arthroplasty. It reflects the patient's assessment of their knee-related health status and benefits of treatment.
EQ-5D-5L | Pre-operative, 1, 2 and 5 years
  EQ-5D-5L is a widely-used patient-administered instrument for describing health-related quality of life
Range of motion (ROM) | Pre-operative, 6 weeks, 3, 12, 24 and 60 months
  ROM will be measured by extension and flexion with a goniometer preoperatively at baseline and at each follow-up visit (6 weeks, 3 months, 12 months, 24 months and 60 months
Kinematic radiostereometric analysis (RSA) | After 12 months
  Knee motion while walking up and down stairs, and during squatting and kneeling activities will be recorded using video fluoroscopy (dynamic RSA) at 12 months.
Plain anterior posterior radiographs and hip, knee and ankle (HKA) radiographs | Pre-operative, 3, 12, 24 and 60 months
  Radiographs obtained for assessment of fixation of the prosthesis and the alignment.
Brief Pain Inventory | Pre-operative, 6 weeks, 3, 12, 24 and 60 months
  We will use three single items to measure worst pain intensity, average pain intensity, and pain interference with walking. Patients rate their pain intensity and pain interference with walking on an 11-point numeric rating scale from 0-10, where 0=no pain/no interference and 10=worst imaginable pain/complete interference.

CONTACTS AND LOCATIONS:
Overall Officials: Arild Aamodt, MD, PhD, Study Director — Lovisenberg Diaconal Hospital, Oslo, Norway
Locations (2):
- Norway (2):
  - Haugesund Rheumatism Hospital, Haugesund
  - Lovisenberg Diaconal Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No